CLINICAL TRIAL: NCT04433104
Title: Allogeneic Human Umbilical Cord-derived Mesenchymal Stem/Stromal Cells for Chronic Obstructive Pulmonary Disease (COPD): Study Protocol for a Matched Case-control, Phase I/II Trial
Brief Title: Umbilical Cord Mesenchymal Stem Cells Transplantation in the Treatment of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VinmecISC1916
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: COPD
Keywords: COPD; umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (UC-MSC trasnplatation) (Experimental): 1 x 10^6 umbilical Cord Mesenchymal Stem Cells per body kg will transplant via the intravenous at baseline, and the second transplantation will be performed 3 months after the first transplantation and combination with Vietnames MOH procedure
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells transplantation; Drug: drug therapy according to Vietnamese MOHS procedure
- control arm (Other): drug therapy according to Vietnamese MOHS procedure
  Interventions: Drug: drug therapy according to Vietnamese MOHS procedure

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells transplantation — Patients assigned to UC-MSC administration groups will receive two administrations at a dose of 1 million cells/kg patient body weight via the IV route with a 3-month intervening interval
  Arms: Treatment (UC-MSC trasnplatation)
Drug: drug therapy according to Vietnamese MOHS procedure — Salbutamol, Terbutaline

SUMMARY:
This trial is to investigate the safety and potential therapeutic efficacy of allogeneic administration of umbilical cord-derived MSCs (UC-MSCs) as a supplementary intervention in combination with standard COPD medication treatments in patients with moderate-to-severe COPD based on the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2019 and Vietnam Ministry of Health's guidelines

DETAILED DESCRIPTION:
The aim of this trial is to investigate the safety and potential therapeutic efficacy of allogeneic administration of umbilical cord-derived MSCs (UC-MSCs) as a supplementary intervention in combination with standard COPD medication treatments in patients with moderate-to-severe COPD based on the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2019 and Vietnam Ministry of Health's guidelines. This matched case-control phase I/II trial is conducted at Vinmec Times City International Hospital, Hanoi, Vietnam between June 2020 and December 2021. In this study, 40 patients will be enrolled and assigned into two age-, gender- and COPD condition-matched groups, including a UC-MSC group and a control group. Both groups will receive standard COPD medication treatment based on the GOLD 2019 guidelines and the Vietnam Ministry of Health protocol. The UC-MSC group will receive two doses of thawed UC-MSC product with an intervention interval of 3 months. The primary outcome measures will include the incidence of prespecified administrationassociated adverse events (AEs) and serious adverse events (SAEs). The efficacy will be evaluated based on the absolute changes in the number of admissions, arterial blood gas analysis, lung function and lung fibrosis via CT scan and chest X-ray. The clinical evaluation will be conducted at baseline and 3, 6, and 12 months post

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD with stage B, C, or D according to GOLD 2019.
* Age between 40-75 years old.
* Both genders.

Exclusion Criteria:

* Smoker or less than 6 months of smoking cessation time.
* Asthma and other pulmonary-related diseases and injuries (including lung tuberculosis, restrictive lung disease, idiopathic pulmonary fibrosis, or lung cancer).
* Acute and/or active infection.
* Cancer.
* Patients with complex cardiovascular diseases (including valvular heart disease, cardiomyopathy, arrhythmia, congenital heart disease, hypertrophy syndrome).
* Liver and kidney failure.
* Pregnancy.
* Patients with life expectancy less than 6 months due to concomitant illness.
* Under immunosuppressive treatment within 8 weeks of the first screening visit.
* Patient diagnosed diabetes with HbA1C>7%

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | up to the 12-month period following treatment
  To assess safety, the number of AEs or SAEs during stem cell administration (72 h) at 3 months, 6 months, and 12 months after discharge will be evaluated

SECONDARY OUTCOMES:
Quality of Life using Georges Respiratory Questionnaire | up to the 12-month period following treatment
  Georges Respiratory Questionnaire has scores range from 0 to 100, with higher scores indicating more limitations
Chest CT | up to the 12-month period following treatment
  Changes of the lung fibrosis on chest CT at 6 months, and 12 months compared with baseline
arterial blood gas analysis (pH) | up to the 12-month period following treatment
  arterial blood gas analysis (pH)
arterial blood gas analysis (PaO2) | up to the 12-month period following treatment
  arterial blood gas analysis (PaO2)
arterial blood gas analysis (PaCO2) | up to the 12-month period following treatment
  arterial blood gas analysis (PaCO2)
arterial blood gas analysis (BE) | up to the 12-month period following treatment
  arterial blood gas analysis (BE)
arterial blood gas analysis (HCO3-) | up to the 12-month period following treatment
  arterial blood gas analysis (HCO3-)
Respiratory functions (FEV1) | up to the 12-month period following treatment
  Respiratory functions (FEV1)
Respiratory functions (FEV1/FVC) | up to the 12-month period following treatment
  Respiratory functions (FEV1/FVC)
Respiratory functions (VC) | up to the 12-month period following treatment
  Respiratory functions (VC)
Respiratory functions (TLC) | up to the 12-month period following treatment
  Respiratory functions (TLC)
Respiratory functions (RV) | up to the 12-month period following treatment
  Respiratory functions (RV)
Respiratory functions (DLCO) | up to the 12-month period following treatment
  Respiratory functions (DLCO)
Respiratory functions (DLNO/DLCO) | up to the 12-month period following treatment
  Respiratory functions (DLNO/DLCO)
inflammatory response (CRP) | up to the 12-month period following treatment
  inflammatory response (CRP)
inflammatory response (Pro-BNP) | up to the 12-month period following treatment
  inflammatory response (Pro-BNP)
inflammatory response (Troponin-T) | up to the 12-month period following treatment
  inflammatory response (Troponin-T)
cytokine analysis from patients' plasma | up to the 12-month period following treatment
  cytokine analysis from patients' plasma
modified medical research council | up to the 12-month period following treatment
  modified medical research council (mMRC)

CONTACTS AND LOCATIONS:
Overall Officials: Duc Minh Hoang, PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec International Hospital Times City, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ribeiro-Paes JT, Bilaqui A, Greco OT, Ruiz MA, Marcelino MY, Stessuk T, de Faria CA, Lago MR. Unicentric study of cell therapy in chronic obstructive pulmonary disease/pulmonary emphysema. Int J Chron Obstruct Pulmon Dis. 2011 Jan 1;6:63-71. doi: 10.2147/COPD.S15292. PMID 21311694
- [Result] Stessuk T, Ruiz MA, Greco OT, Bilaqui A, Ribeiro-Paes MJ, Ribeiro-Paes JT. Phase I clinical trial of cell therapy in patients with advanced chronic obstructive pulmonary disease: follow-up of up to 3 years. Rev Bras Hematol Hemoter. 2013;35(5):352-7. doi: 10.5581/1516-8484.20130113. PMID 24255620
- [Result] Stolk J, Broekman W, Mauad T, Zwaginga JJ, Roelofs H, Fibbe WE, Oostendorp J, Bajema I, Versteegh MI, Taube C, Hiemstra PS. A phase I study for intravenous autologous mesenchymal stromal cell administration to patients with severe emphysema. QJM. 2016 May;109(5):331-6. doi: 10.1093/qjmed/hcw001. Epub 2016 Jan 27. PMID 26819296
- [Derived] Hoang DM, Nguyen KT, Nguyen AH, Nguyen BN, Nguyen LT. Allogeneic human umbilical cord-derived mesenchymal stem/stromal cells for chronic obstructive pulmonary disease (COPD): study protocol for a matched case-control, phase I/II trial. BMJ Open. 2021 May 13;11(5):e045788. doi: 10.1136/bmjopen-2020-045788. PMID 33986057